CLINICAL TRIAL: NCT06513871
Title: Evaluating the Impact of Community-Based Mindfulness and Musical Programs on Psychiatric Measures, Social Perception Tasks 2d.
Brief Title: Evaluating Social Perception Dynamics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000028866_d; 2R25MH071584-11 (NIH)
Record Dates: First submitted 2024-07-10; First posted 2024-07-22 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Mental Health Issue; COVID-19
Keywords: Mindfulness; Meditation; Music
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Component 2d. Social Perception Tasks (Experimental): Participants will take part in social perception tasks in speed-dating like interactions with individuals in which they are not allowed to verbally communicate. After silently interacting with each partner, subjects will be prompted to answer survey questions about their perceptions of their partner and their interaction. This task will take place in a variety of settings.
  Interventions: Behavioral: Social perception tasks

INTERVENTIONS:
Behavioral: Social perception tasks — social perception tasks

SUMMARY:
Mental health vulnerability due to stress is increased in People of African Descent (PADs) in America due to disproportionate effects of racism, poverty, education, and criminal justice sentencing. Various meditation and mindfulness approaches have provided evidence of measured reductions in multiple negative dimensions of stress. However, the majority of these studies do not have an adequate representation of PADs or other marginalized groups and are not designed to be culturally relevant or community based. Music has been shown to alleviate multiple symptoms of stress and has been shown to be a preferred and effective support for meditation and mindfulness. However, its role in stress management in PADs engaged in meditation or mindfulness is seldom studied. This study aims to evaluate the effects of a virtual, community-based music mindfulness program on stress management in PAD community members with anxiety and depression during COVID19.

Component 2d. Social Perception Tasks: Participants may be asked to take part in social perception tasks in which they will be asked to indicate their social perception and connection felt with various partners.

DETAILED DESCRIPTION:
The investigators also propose a study to investigate the effects of communal drumming in reducing anxiety and increasing connectedness within drum circle community. Investigators hypothesize that these intervention will lead to reductions in scores on stress scales and will provide preliminary data for studies evaluating these types of community programs as an adjunct to the standard of care.

Paradigms will be designed such that participants experience speed-dating like interactions with individuals in which they are not allowed to verbally communicate. After silently interacting with each partner, subjects will be prompted to answer survey questions about their perceptions of their partner and their interaction. This task will take place in a variety of settings.

This task was developed to quantify group dynamics. Participants that are enrolled and consented in a study are given a participant ID number. Each participant sits 2 feet across from another participant. They are paired with that participant for 30 seconds. They are instructed that they can look freely across at their own will. After 30 seconds they are asked to answer the following questions on a Likert scale 1-7 about the interaction with the other participant:

What is your partner's ID? How connected do you feel to this partner? (very unconnected-very connected) How approachable do you think this person is? (very unapproachable-very approachable) How likely is this person to be in your socioeconomic class? (very unlikely-very likely) How likely is this person to share your political views? (very unlikely-very likely) How willing are you to discuss a controversial subject with this partner? (very unwilling - very willing) How willing are you to compromise to solve a complex problem with this partner? (very unwilling - very willing)

Following this they are paired with another participant in the group and complete the same questions. This continues until they have been matched with all other participants.

ELIGIBILITY:
Inclusion Criteria:

* ages 16 and older

Exclusion Criteria:

* ages 15 and younger

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Mean score individual subjective rating of social connection during session | baseline on day of study and 5 minutes after intervention
  Rating of subjective connectedness will be assessed using a Likert scale with total score range from 1-5, with higher scores indicating more connectedness.

SECONDARY OUTCOMES:
Mean score group subjective rating of social connection post session | baseline on day of study and 5 minutes after intervention
  Rating of subjective connectedness will be assessed using a Likert scale with total score range from 1-5, with higher scores indicating more connectedness.

CONTACTS AND LOCATIONS:
Overall Officials: AZA Allsop, MD, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - BLOOM, New Haven, Connecticut
  - Musical Intervention Studios, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
De-identified, aggregate data will be shared through pre-prints, publications, and community town hall meetings.